CLINICAL TRIAL: NCT01823822
Title: Influence of Protein Supplements on Serum Insulin-like Growth Factor-I Levels in Women With Anorexia Nervosa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Rene Rizzoli, René Rizzoli, MD (Principal Investigator), University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-182; NU185 (Other: Danone Research)
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Protein supplements; IGF-I
MeSH Terms: conditions — Anorexia Nervosa | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral protein supplement (Tested product) (Experimental)
  Interventions: Dietary Supplement: Oral protein supplement (Tested product)
- Iso-caloric supplement (Control product) (Active Comparator)
  Interventions: Dietary Supplement: Iso-caloric supplement (Control product)

INTERVENTIONS:
Dietary Supplement: Oral protein supplement (Tested product) — Test product: oral protein supplement, sweetened flavoured dairy product, type fresh cheese rich in milk protein (15 g/150 grams). Dosage is 2 pots daily, at least 5 days/week for 4 consecutive weeks.
  Arms: Oral protein supplement (Tested product)
Dietary Supplement: Iso-caloric supplement (Control product) — Control product: sweetened flavoured fresh cheese, with low milk protein content (3 g/150 grams). Dosage is 2 pots daily, at least 5 days/week for 4 consecutive weeks.
  Arms: Iso-caloric supplement (Control product)

SUMMARY:
This multicentre, randomised, double-blind, 2-parallel group, controlled trial aims to investigate whether oral milk protein supplements led to increase in serum Insulin-like Growth Factor-I levels (IGF-I) as compared with a control group fed with an iso-caloric supplement, in women with anorexia nervosa. Subjects receive either 150g/day of tested product or control product for 4-week, followed by a 4-week follow-up.

DETAILED DESCRIPTION:
Study centres: 4 active centres in France and 2 active centres in Switzerland

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 to 40 years (bounds included).
* Women with a serum IGF-I level below the 25th percentile of the reference value according to the age (bounds included).
* Women who had given written inform consent.
* Women with DSM-IV-confirmed anorexia nervosa lasting for at least 6 months. Women with concomitant binge eating and purging type are also included.
* Women admitted in-hospital for weight and nutritional rehabilitation. It is anticipated that the patient will stay in-hospital during the full duration of the 4-week supplementation phase, and at least 5 weeks within the study.
* Women being already regular consumers of dairy products.
* For women with childbearing potential, use of a contraceptive method.
* Discontinuation of any mineral and vitamin supplements containing calcium and vitamin D, 1 week before starting the product consumption and during the study.

Exclusion Criteria:

* Women with primary amenorrhea;
* Women with lactose intolerance;
* Women with any other metabolic disease that could affect bone metabolism: osteogenesis imperfecta, Paget's disease of bone, hyperthyroidism, primary hyperparathyroidism;
* Women with current or past neoplasm;
* Women with any other severe comorbidity;
* Pregnant or breast feeding women;
* Women with epilepsy;
* Women with any current or past use of the following treatments: bisphosphonates, calcitonin, steroids;
* Patients enrolled in another clinical study within the last 4 weeks;
* Patients having already received oral nutritional supplements or who need to receive other oral or intravenous (IV) supplements during the follow-up;
* Patients having received oral or IV nutritional supplements within two weeks before the inclusion;
* Patients having willed to participate in another clinical study during the present study phase and 4 weeks after the end of their participation in the present study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Serum insulin like growth factor-1 (IGF-I) level | 4-week
  The main study product effect criterion is the IGF-I level over the 4-week consumption period.

CONTACTS AND LOCATIONS:
Overall Officials: René Rizzoli, MD, Principal Investigator — Bone Diseases Service, Department of Internal Medicine Specialties, University Hospitals and Faculty of Medicine of Geneva
Locations (1):
- Bone Diseases Service, Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Trombetti A, Carrier E, Perroud A, Lang F, Herrmann FR, Rizzoli R. Influence of a fermented protein-fortified dairy product on serum insulin-like growth factor-I in women with anorexia nervosa: A randomized controlled trial. Clin Nutr. 2016 Oct;35(5):1032-8. doi: 10.1016/j.clnu.2015.10.014. Epub 2015 Nov 5. PMID 26602423